CLINICAL TRIAL: NCT04619056
Title: First-in-man Clinical Trial to Assess Safety and Tolerability of CEB-01 PLGA Membrane in Patients With Recurrent or Locally Advanced Retroperitoneal Soft Tissue Sarcoma After Surgery
Brief Title: First-in-man Clinical Trial of CEB-01 PLGA Membrane in Recurrent or Locally Advanced Retroperitoneal Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CEBIOTEX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEB-01-RLS01-CT; 2018-001026-25 (EudraCT Number)
Record Dates: First submitted 2020-10-30; First posted 2020-11-06 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Soft Tissue Sarcoma; Recurrent Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Retroperitoneal; Recurrent or locally advanced; CEB-01 PLGA membrane; SN-38; Local drug delivery system
MeSH Terms: conditions — Sarcoma; Recurrence | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: This is an open label, first-in-human clinical trial that will be conducted in 3 dose-escalation cohorts (3-6 patients each) and in an expansion cohort, at the highest dose determined to be safe and tolerable.
  CEB-01 loaded with a SN-38 dose between 9 and 36 mg will be allocated to each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): CEB-01 with total SN-38 dose: 9 mg
  Interventions: Drug: CEB-01 membrane loaded with SN-38
- Cohort 2 (Experimental): CEB-01 with total SN-38 dose: 18 mg
  Interventions: Drug: CEB-01 membrane loaded with SN-38
- Cohort 3 (Experimental): CEB-01 with total SN-38 dose: 36 mg
  Interventions: Drug: CEB-01 membrane loaded with SN-38

INTERVENTIONS:
Drug: CEB-01 membrane loaded with SN-38 — CEB-01 is a polymeric drug with a delivery system loaded with SN-38, and will be placed in the surgical bed at the time of tumor resection.

SUMMARY:
This is an open label, first-in-man clinical trial to assess safety and tolerability of CEB-01 PLGA membrane in patients with recurrent or locally advanced retroperitoneal soft tissue sarcoma after surgery.

The trial will be conducted in 3 dose-escalation cohorts (3 patients each, enrolling patients one by one, after 4 weeks of observation and agreement of Scientific Committee and DMC) and in an expansion cohort, using the highest safe and tolerable dose. The study will follow a 3+3 modified design; dose escalation will follow a modified Fibonacci method. CEB-01 carrying a SN-38 dose between 9 and 36 mg will be placed in the surgical bed at the time of tumor resection.

DETAILED DESCRIPTION:
CEB-01 is a poly(lactic-co-glycolic acid) (PLGA) polymeric drug with a delivery system loaded with SN-38, and will be placed in the surgical bed at the time of tumor resection.

CEB-01 carrying a SN-38 dose between 9 and 36 mg will be administered. CEB-01 will be placed on all surfaces that were in contact with and/or were infiltrated by the tumor.

Confirmatory central reviewing of diagnosis will be performed for all patients, using tumor samples obtained during surgery; additionally, patients will also be included according to local Pathological Anatomy (PA) diagnosis.

Patients will be followed-up once every week during the first 8 weeks of the study, and then every 2 weeks up to 12 weeks after implantation of CEB-01. Thereafter, follow-up schedule will be as per normal practice until study completion.

Efficacy assessment will be performed by Magnetic Resonance Imaging (MRI) [Computed tomography (CT) scan and Positron Emission Tomography (PET-CT) are also allowed] according to RECIST 1.1 criteria. Baseline image determination will be performed at week 12 (±3 days) after surgery; if the image analysis is not conclusive due to wound healing in the tumor bed, it will be repeated on week 16 (±3 days) post-surgery, and every 12 weeks thereafter.

A pharmacokinetic assessment of SN-38 will be performed in all patients, and the Cmax, Tmax, half-life, and area under the time-drug concentration curve (AUC) of the drug will be determined. Blood samples will be collected at baseline and at 8 time points after CEB-01 implantation.

Assessment of adverse events, safety, and toxicity will be performed according to the Common Terminology Criteria for Adverse Events (CTCAE - version 5.0) at each patient visit from the time of Informed Consent until the end of the study.

Quality of Life based on EORTC Quality of Life Questionnaire (QLQ) 30 will be measured prior surgery, at month 1 and month 3.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Histologically confirmed diagnosis of locally advanced (T3 -T4, American Joint Committee on Cancer (AJCC)/primary tumor, regional lymph nodes, and distant metastases staging system (TMN) 8th Edition) and/or relapsed (any) retroperitoneal soft tissue sarcoma (liposarcoma, leiomyosarcoma, a solitary fibrous tumor (SFT), pleomorphic sarcoma, or a malignant nerve sheath tumor). Patients with local advanced (T3 -T4,AJCC/TMN 8th Edition) and/or relapse and metastatic disease who are candidates for local surgery without option of systemic treatment, are also eligible for the trial.
3. Pathology specimens available for centralized review. Submission of formalin-fixed paraffin-embedded (FFPE) tumor tissue for central reviewing is required; if a FFPE block cannot be provided, then 10 unstained, positively-charged slides of 4-5 um thickness must be submitted.
4. Size of tumor (visible or previously inadequately resected) >5 cm at instrumental staging (CT, MRI).
5. Normal liver, renal, hematological, and cardiac function as defined by biochemical and hematological parameters as follows: Hb >11 g/dL, platelets >100.000/mm3, White Blood Cells (WBC) >3000/mm3, neutrophil count >1500/mm3, albumin >3.0 g/dl, Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) <2.5 times the upper limit of normality (ULN), bilirubin <2 times the ULN, creatinine <1.5 mg/dl or creatinine clearance > 60 ml/min.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status <2.
7. No concomitant radiotherapy or chemotherapy planned.
8. Life expectancy greater than 6 months.
9. Female subjects of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at time of screening.
10. Men and women of childbearing potential must be willing to use adequate contraception throughout the study and for 3 months after surgery.
11. Ability to understand and the willingness to sign a written informed consent document; subject has signed an Informed Consent Form (ICF) prior to any screening procedures and is able to comply with protocol requirements.

Exclusion Criteria:

1. Pregnancy or lactation. Note: Pregnant women are excluded from this study; if the patient is a lactating mother, breastfeeding should be discontinued.
2. Other malignancies within past 5 years, with the exception of carcinoma in situ of cervix and basocellular skin cancers treated with eradicating intent.
3. Serious psychiatric disease that precludes informed consent or limits compliance
4. Medical condition limiting survival to less than 6 months.
5. Uncontrolled bacterial, viral or fungal infection.
6. Active viral hepatitis or chronic liver disease.
7. Impossibility of ensuring adequate follow-up.
8. Contraindication to magnetic resonance imaging (MRI), including presence of a pacemaker or an aneurysm clip, severe claustrophobia, a known reaction to the gadolinium contrast dye, or body weight that could interfere with the feasibility of a MRI.
9. Major surgery within 14 days prior to starting study drug or still in recovery after experiencing surgical complications; neither tumor biopsy nor central line insertion are considered a major surgery.
10. Unable or unwilling to stop the use of herbal supplements; the use of nutritional supplements may be allowed after review by a study pharmacist to confirm no significant risk of interaction with eribulin or radiation.
11. Other relevant concomitant illnesses.
12. Patients previously treated with Irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Recommended Doses for Phase II (Maximum tolerated dose) | Through 2 weeks
  The number of patients experiencing dose limiting toxicities during the Dose Limiting Toxicities (DLT) observation period of 2 weeks.

SECONDARY OUTCOMES:
Frequency of Adverse Events (AEs) (Safety) | Through study completion, average 2 years
  Frequency of adverse events reported classified by type and severity.
Frequency of Treatment Related Adverse Events (TRAEs) (Toxicity) | Through study completion, average 2 years
  Frequency of treatment related adverse events reported classified by type and severity.
Time to local relapse (TTLR) | Through study completion, average 2 years
  Time from the start of treatment to the date of local relapse according to the RECIST 1.1 criteria, or death due to any cause. Those patients who are alive and have not relapsed at the last follow-up, will be censored at the date of the last follow-up.
  Relapse definition: For patients in which R0 is obtained by surgery, relapsed should be considered when disease reappears with size > 1 cm (measurable disease). For patients with R1 or R2, RECIST 1.1 guideline should be used for disease progression definition.
Progression Free Survival (PFS) | Through study completion, average 2 years
  Time from the start of treatment to the date of the first progression according to the RECIST 1.1 criteria, or death due to any cause. Those patients who are alive and have not progressed at the last follow-up, date of progression will be censored at the date of the last follow-up.
Overall Survival (OS)(until 24 months of Follow Up (FU)) | Through study completion, average 2 years
  Median of overall survival. Time from the start of the trial treatment to the date of exitus for any cause. In those patients who are alive at the last follow-up, OS will be censored by the date of the last follow-up in which the patient was alive.
Quality of life: EORTC QLQ 30 | Prior to surgery, at month 1 and month 3 after surgery
  Questionnaire developed and validated to assess the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Sebio, M.D. Ph.D., Study Chair — Hospital Universitari de la Santa Creu i Sant Pau
Locations (5):
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No